CLINICAL TRIAL: NCT04723277
Title: TeaLeaF: Teachers Leading the Frontlines
Brief Title: Efficacy of Teacher-delivered Child Mental Healthcare in Primary Schools of India
Acronym: TeaLeaF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of North Bengal, India (Unknown); Darjeeling Ladenla Road Prerna (Unknown); Broadleaf Health and Education Alliance (Other); University of Colorado, Denver (Other); American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-2868
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Child Behavior Disorders
Keywords: child; child behavior; child behavior disorders; global health; India; mental health; schools; school mental health services; school teachers/psychology; students/psychology
MeSH Terms: conditions — Child Behavior Disorders; Child Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a stepped-wedge cluster randomized trial. Given the nature of the intervention, each school will be a cluster and each step will be an academic year. Randomization will occur at the school level. All schools will initially receive the control condition (EUC) and will be randomly and sequentially transitioned into the intervention arm. A qualitative exploration of context and process will be embedded within the framework of the randomized control trial. An embedded approach has been chosen to facilitate a high level of integration between the qualitative and quantitative components of the study.
Who Masked: Outcomes Assessor
Masking Description: Complete double-blinding is not possible in this mental health intervention trial as trial participants and the intervention team will be aware of their status. However, to minimize bias and the risk of unmasking, the field team will be separated into intervention and data collection teams. The data collection team will be blinded to intervention allocation at the cluster-level and treatment status at the individual child level. Additionally, while over time it may be likely that children and caregivers are aware of the intervention delivered, they will not be explicitly informed of this allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tealeaf - Year 1: Clusters (schools) and associated participants assigned to sequence 1 (Experimental): Clusters (schools) and associated participants assigned to sequence 1 will be under the EUC condition in the 1st year of trial participation and under the Tealeaf condition in all subsequent years.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- Enhanced Usual Care - Year 1: Clusters (schools) and associated participants assigned to sequence 2 (Active Comparator): Clusters (schools) and associated participants assigned to sequence 2 will be under the EUC condition in the 1st and 2nd year of trial participation and under the Tealeaf condition in all subsequent years.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- Tealeaf - Year 2: Clusters (schools) and associated participants assigned to sequence 1 (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family.
  Interventions: Behavioral: Tealeaf-Mansik Swasta (Tealeaf)
- Enhanced Usual Care - Year 2: Clusters (schools) and associated participants assigned to sequence 2 (Active Comparator): EUC (control arm)
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- Tealeaf - Year 3: Clusters (schools) and associated participants assigned to sequence 1 (Experimental): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family.
  Interventions: Behavioral: Tealeaf-Mansik Swasta (Tealeaf)
- Enhanced Usual Care - Year 3: Clusters (schools) and associated participants assigned to sequence 2 (Active Comparator): Active intervention: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family.
  Interventions: Behavioral: Tealeaf-Mansik Swasta (Tealeaf)

INTERVENTIONS:
Behavioral: Tealeaf-Mansik Swasta (Tealeaf) — Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Mental health challenges are understood through basic functional behavior assessments, providing a framework for the analysis of observable behaviors. Teachers deliver care primarily through the incorporation of basic therapeutic interactions into classroom instruction time, supplemented by one-on-one interactions with the child and family. Teachers receive ongoing supervision and support from the intervention team including monthly site visits supplemented by monthly and as-needed telephone discussions.
  Arms: Enhanced Usual Care - Year 3: Clusters (schools) and associated participants assigned to sequence 2; Tealeaf - Year 2: Clusters (schools) and associated participants assigned to sequence 1; Tealeaf - Year 3: Clusters (schools) and associated participants assigned to sequence 1
Behavioral: Enhanced Usual Care (EUC) — Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment.
  Arms: Enhanced Usual Care - Year 1: Clusters (schools) and associated participants assigned to sequence 2; Enhanced Usual Care - Year 2: Clusters (schools) and associated participants assigned to sequence 2; Tealeaf - Year 1: Clusters (schools) and associated participants assigned to sequence 1

SUMMARY:
Twenty percent of all children struggle with mental health challenges, most of whom will remain unrecognized, unsupported, and unable to access quality care. A major barrier to closing this care gap is a lack of evidence-based delivery models that are contextualized to low-resource settings. The aim of this study is to evaluate the efficacy of teacher-delivered transdiagnostic mental healthcare for children in rural primary schools of India. Implementation process and context will also be examined.

This is a stepped-wedge cluster randomized controlled trials (SW-CRCT), with an embedded qualitative evaluation, that will be conducted in low-cost private primary schools in the rural Darjeeling Himalayas of India.

The primary outcome is children's mental health status measured by the Achenbach System of Empirically Based Assessment (ASEBA) Teacher Report Form and Strengths and Difficulties Questionnaire. Secondary outcomes include: 1) daily functioning measured by the Adaptive Behavior Assessment System (ABAS-3), 2) academic achievement measured by the Annual Status of Education Report (ASER) tool, and 3) school attendance. Outcome data will be collected at baseline and endline in each academic year. The primary analysis for each outcome is the mean score at endline for children receiving targeted intervention (Tealeaf: Mansik Swastha or Enhanced Usual Care) between trial arms. The primary hypothesis is that children receiving mental health struggles receiving the Tealeaf intervention will demonstrate improved mental health compared to children with mental health struggles receiving enhanced usual care.

The goal of the embedded qualitative study will be to explore the effect of cultural and social context on intervention implementation and efficacy, how and why changes may occur, and the culture, context, and community in which the study occurs. This qualitative research will be driven by the scientific standard of advanced qualitative methods (ethnography and participant observation).

This trial may offer a new approach to caring for children with mental health struggles that is potentially scalable in India as it empowers existing classroom teachers.

DETAILED DESCRIPTION:
Expanding access to children's mental health care is a critically important global health challenge. There is a substantial gap between who would benefit and those who receive care. Task-shifting has been one widely used approach to closing care gaps for other health challenges. However, alternative models for mental health care delivery targeting school-aged children, including task-shifting, are rare. Classroom teachers are uniquely positioned to deliver children's mental health care in a transdiagnostic task-shifting model.

TeaLeaf (TEAchers LEAding the Frontlines) is a research program based in the Darjeeling Himalayas with the goal to develop, test, and scale alternative and combined models of education and mental health care that leverage classroom teachers and synergies between the fields of education and child psychiatry to improve the lives of children with mental health struggles. A novel mental health program (Tealeaf-Mansik Swastha) has been developed with the aims to (i) improve access to evidence-based mental healthcare for children, (ii) improve children's mental health outcomes, and (iii) improve children's wellbeing, development, and academic functioning. Through this intervention teachers are empowered to incorporate simple, easy-to-use yet evidence-based mental health techniques in their everyday interaction with targeted students. This model shifts the paradigm of care from difficult to access episodic intervention to ongoing, therapeutic interactions occurring through their day.

Formative and pilot studies have demonstrated that teachers can deliver evidence-based mental health care with fidelity, and that this approach is broadly acceptable to stakeholders, and an early signal for effectiveness. In the present study, an evaluation of efficacy will be coupled with an embedded qualitative exploration of context and process. Evaluating efficacy, implementation processes of the program, and the context in which it occurs will generate valuable insights into how children's mental health care can best be delivered in resource-limited settings.

The primary objective of the study is to evaluate the efficacy of teacher-delivered transdiagnostic mental healthcare for school-aged children in resource-limited primary schools. The primary hypothesis is that children receiving the Tealeaf intervention will demonstrate improved mental health compared to children receiving Enhanced Usual Care (EUC). Secondary objectives are: 1) to evaluate the efficacy of the intervention with regards to children's daily functioning, academic achievement, and school attendance; 2) to explore the influence of culture and social context on intervention implementation and efficacy; 3) to evaluate implementation processes in order to understand how and why change may occur; and 4) to explore the locatedness of the site of intervention within the larger historical and socio-cultural context.

The study will be conducted as a SW-CRCT. Within the four-year TeaLeaF trial, a prospective 3-year sub-study has been defined. The original protocol was modified to include this sub-study [TeaLeaF(+); registered at Clinical Trials Registry - India (CTR-T)] due to the emergence of the COVID-19 pandemic. TeaLeaF(+) is a 3-year SW-CRCT with a similar structure and analysis plan to TeaLeaF but prospectively defined to begin in 2021. This sub-study will facilitate adjustment in the light of many changes in the broader context arising as a result of the impact of the COVID-19 pandemic and associated school closure.

The study setting is the rural Darjeeling Himalayas, a region of the state of West Bengal in India. The primary site of the intervention will be rural, low-cost community private schools. Low-cost private schools (rather than government schools) were chosen for this study because 1) this is the setting where the highest proportion of children in rural Darjeeling are educated, 2) implementation is more likely to occur with fidelity and quality in this setting, and 3) this setting represents a better environment for assessment of intervention efficacy.

The analysis for the primary outcome (mental health status) and secondary outcomes (daily functioning, academic achievement, and school attendance) will be conducted as a comparison between the intervention arm (Tealeaf) and control arm (EUC) within the context of the stepped wedge framework. The primary analysis will be based on child-level data for children receiving targeted intervention and will be a comparison of mean scores at endline.

A secondary analysis, utilizing a similar approach will be conducted to compare outcomes among a representative subsample of children not selected for targeted intervention between trial arms. An additional secondary analysis will be used to compare children selected to receive intervention with this representative subsample within each trial arm.

Additional analyses will be conducted for the following pre-specified subgroups: 1) gender/sex, 2) age (<=; >=8 years old) and 3) baseline mental health status. The investigators will also conduct a series of pre-specified exploratory analysis on sub-scales or domains for the main outcome measures. A cost-analysis will be performed to estimate the resources required to deliver Tealeaf and EUC.

All analysis will be conducted for both the 4-year TeaLeaF trial and the 3-year post-COVID sub-study [Tealeaf(+)]

The overarching goals of the embedded qualitative study will be to explore the effect of cultural and social context on intervention implementation and efficacy, how and why changes, may occur, and the culture, context, and community in which the study occurs. Grounded research techniques will be used to understand the participant's views and experiences in their context and to shed light on how 'process' aspects of the Tealeaf intervention are impacting communities, teachers, children, and families in a specific cultural context.

To that effect, the qualitative research will not be based on hypothesis testing. Rather it will be driven by the scientific standards of advanced qualitative methods (ethnography and participant observation) where iterative learning and reflection drive data collection and analysis. For this research, a subsample of schools will be selected through stratified purposive sampling. Within each school, in-depth longitudinal direct observation and interviews (and as needed focus groups) with school principals, teachers, parents, caregivers, and children enrolled in the study. This will be supplemented with field notes, process documentation, and data arising from project monitoring.

This trial is the first to evaluate the efficacy of teacher-delivered transdiagnostic mental healthcare for school-aged children in primary schools of a low-to-middle income county. The results of this study are expected to contribute to the limited evidence base for alternative models of children's mental health care in low-resource settings.

During the first year of the trial (2021), the study team will only use the first primary outcome measure, Mean Difference on the Achenbach System of Empirically Based Assessment (ASEBA) Teacher Report Form Total Problem Scale for the following reasons:

1. There is no control group to compare against
2. There is no EUC condition
3. During the 2021 year, we are most interested in identifying any confounding of primary outcome during COVID

ELIGIBILITY:
Inclusion Criteria:

Schools:

* Does not receive government aid (i.e., not subject to the rules and regulations of government or government-aided schools
* At least 3 full-time classroom teachers on staff
* Annual student fees $180/11,500 Indian rupee (INR) or less

Teachers:

* Employed at a participating school
* Have primary teaching responsibility in the primary grade level
* Are 18 years or older
* Children
* Enrolled in class I-IV
* Enrolled in the classroom of a participating teacher

Exclusion Criteria:

Schools:

* Not located in the rural Darjeeling Himalayas (defined as the Mirik, Kurseong, and Darjeeling Sadar sub-divisions of the Darjeeling District and outside the statutory towns of Darjeeling, Kurseon, and MIrik)

Teachers

* Have been convicted and/or are under investigation for any child-related misconduct or maltreatment.

Children:

* Do not have a parent or guardian who can provide informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Difference on the Achenbach System of Empirically Based Assessment (ASEBA) Teacher Report Form Total Problem Scale | 8 months from baseline
  ASEBA Teacher Report Form (TRF) Total Problems Scale is a standardized tool to assess health challenges in children. A raw score is derived by summing responses to 113 problem behavior questions with responses scored from 0 to 2. Higher scores indicate greater problem severity. This raw score is converted into T-scores, and children with Total Problem Scale t-scores lower than 60 are classified in the normal group, children with scores ranging from 60-63 are classified as borderline, and children with scores above 63 were classified as clinical.
Mean Difference at Endline on the Strengths and Difficulties Questionnaire Total Difficulties Score | 8 months from baseline
  The Strengths and Difficulties Questionnaire Total is a standardized tool to measure for psychopathology in children and adolescents. A Total Difficulties scale score is derived by summing items from four problem subscales (emotional, conduct, hyperactivity/inattention, and peer relationship), while a fifth subscale (prosocial functioning) does not contribute to the overall severity score. Scores also include an internalizing score, externalizing score, and impact score. Individual problem scale items are scored from 0 to 2 (with higher scores indicating greater problem severity).

SECONDARY OUTCOMES:
Mean Difference on Global Adaptive Composite Score of a locally-contextualized version of the Adaptive Behavior Assessment System 3rd Edition (ABAS-3). | 8 months from baseline
  The ABAS-3 measures 11 essential daily functioning skill areas (communication (raw score range (RSR) 0-66), community use (RSR 0-45), functional academics (RSR 0-66), health and safety ( RSR 0-45), home or school living (RSR 0-66), leisure (RSR 0-48), self-care (RSR 0-57), self-direction (RSR 0-63), social (RSR 0-66), and work (RSR 0-57)) within 3 major adaptive domains (Conceptual (RSR 0-195), Social (RSR 0-114), and Practical (RSR 0-213)) for students age 5-21 years. On a 4-point response scale (range 0-3), raters indicate whether, and how frequently, the individual performs each activity. A Global Adaptive Composite (GAC) score is derived from standardizing the sum of scores from all skill areas except work. The GAC is standardized to a mean of 100 with a standard deviation of 15, with the standardized sum ranging from a minimum category of "70 or less" and a maximum category of "130 or greater". A higher score indicates higher daily functioning skills in the included areas.
Mean Difference on Annual Status of Education Report (ASER) Composite Score | 8 months from baseline
  The ASER is a measure of academic performance of children 6-14 in India. Domains assessed include reading, math, and English. The tool was expanded to include assessment of higher-order functions. A composite score is derived from the score on individual assessment domains. The ranges for each domain are as follows: Math (0-10), Reading (0-5), Total (0-15). A higher score indicated that the child scored at a higher grade level.
Mean Difference in Proportion of School Days Absent | 8 months from baseline
  School attendance data will be obtained from teacher-completed and school-maintained log books of student attendance. Given that the school year varies by school, the number of days a child is absent will be converted to a proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cruz, MD, EdM, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- DLR Prerna, Darjeeling, West Bengal, India

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) generated during and/or analyzed during the study will not be publicly available due to the potential for deductive disclosure but may be available from Darjeeling Ladenla Road (DLR) Prerna on reasonable request.

REFERENCES:
- [Background] Tealeaf: Mansik Swastha [Internet]. @TeleafMansikSwastha. [cited 2020 Oct 8]. Available from: https://www.facebook.com/TealeafMansikSwastha
- [Background] Global Child Mental Health Collaborative: creating, testing, and implementing alternative systems of child and adolescent mental health care. [Internet]. [cited 2020 Oct 7]. Available from: https://globalchildmentalhealth.web.unc.edu/
- [Derived] Giri P, Lamb MM, Fuentes VC, Thapa A, Bhattarai S, Dukpa C, Shrestha CC, Ekhteraei S, Vanderburg JL, Windsor B, Rauniyar AK, Hampanda K, Gaynes BN, Lama R, Matergia M, Cruz CM. Comparative child mental health and academic outcomes after primary school teachers deliver task-shifted mental health care in India. Discov Ment Health. 2025 Jun 18;5(1):90. doi: 10.1007/s44192-025-00217-2. PMID 40531254